CLINICAL TRIAL: NCT02180256
Title: Effect of Endometrial Scratching on Assisted Reproduction Outcomes: a Randomized Controlled Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The main investigators are no longer working at the the center
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Wellington P Martins, MD, Researcher, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CAAE: 30504514.6.0000.5440
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Subfertility
Keywords: IVF; ICSI; Embryo transfer; Assisted reproduction; Endometrial injury; Endometrial scratching
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Endoscratching, non-RIF (Experimental): Endometrial scratching. Women with no more than 1 previous unsuccessful embryo transfer. Pipelle in the first seven days of the menstrual cycle, just before starting controlled ovarian stimulation.
  Interventions: Procedure: Endometrial Scratching
- Control, non-RIF (No Intervention): No intervention. Women with no more than 1 previous unsuccessful embryo transfer.
- Endoscratching, RIF (Experimental): Endometrial scratching. Women with 2 or more previous unsuccessful embryo transfers. Pipelle in the first seven days of the menstrual cycle, just before starting controlled ovarian stimulation.
  Interventions: Procedure: Endometrial Scratching
- Control, RIF (No Intervention): No intervention. Women with 2 or more previous unsuccessful embryo transfers.

INTERVENTIONS:
Procedure: Endometrial Scratching — The intentional damage to the endometrium performed with the objective of improving the reproductive outcomes of women desiring pregnancy.
  Other Names: Endometrial injury; Endometrial biopsy; Endoscratching
  Arms: Endoscratching, RIF; Endoscratching, non-RIF

SUMMARY:
To examine whether endometrial scratching (or injury) using a Pipelle endometrial sampler, performed on the first seven days of the menstrual cycle, is able to improve pregnancy rates in women who will be submitted to a fresh embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* First four days of the menstrual cycle, just before starting controlled ovarian stimulation for planned IVF and fresh embryo transfer.
* Not have performed endometrial scratching in the last 90 days.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Live birth | 1 year
  The number of participants who delivered a living baby in each arm. The denominator will be the number of women randomized to each arm. This outcome will be assessed by examining the medical records and telephone contact.

SECONDARY OUTCOMES:
Clinical pregnancy | 8 weeks
  The number of participants achieved clinical pregnancy detected by ultrasound (either intrauterine or ectopic). The denominator will be the number of women randomized to each arm. This outcome will be assessed by examining the medical records and telephone contact.
Miscarriage | 20 weeks
  The number of participants who experienced spontaneous loss of a clinical pregnancy before 20 completed weeks of gestational age. The denominator will be the number of women who achieved clinical pregnancy in each arm. This outcome will be assessed by examining the medical records and telephone contact.
Multiple pregnancy | 8 weeks
  The number of pregnant participants with more than one gestational sac (twins/triplets). The denominator will be the number of women who achieved clinical pregnancy in each arm. This outcome will be assessed by examining the medical records and telephone contact.

OTHER OUTCOMES:
Implantation rate | 8 weeks
  The number of gestational sacs divided by the number of transferred embryos in each arm. This outcome will be assessed by examining the medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Wellington P Martins, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hc-Fmrp-Usp, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Nastri CO, Teixeira DM, Ferriani RA, Martins WP. The overlooked endometrial injury underlying hysteroscopy procedures. Reprod Biomed Online. 2014 Jul;29(1):140. doi: 10.1016/j.rbmo.2014.03.021. Epub 2014 Apr 28. No abstract available. PMID 24835342
- [Background] Nastri CO, Ferriani RA, Raine-Fenning N, Martins WP. Endometrial scratching performed in the non-transfer cycle and outcome of assisted reproduction: a randomized controlled trial. Ultrasound Obstet Gynecol. 2013 Oct;42(4):375-82. doi: 10.1002/uog.12539. Epub 2013 Sep 2. PMID 23754314
- [Background] Nastri CO, Teixeira DM, Martins WP. Endometrial injury in the menstrual cycle prior to assisted reproduction techniques to improve reproductive outcomes. Gynecol Endocrinol. 2013 May;29(5):401-2. doi: 10.3109/09513590.2012.760193. Epub 2013 Jan 22. No abstract available. PMID 23339704
- [Background] Nastri CO, Gibreel A, Raine-Fenning N, Maheshwari A, Ferriani RA, Bhattacharya S, Martins WP. Endometrial injury in women undergoing assisted reproductive techniques. Cochrane Database Syst Rev. 2012 Jul 11;(7):CD009517. doi: 10.1002/14651858.CD009517.pub2. PMID 22786529